CLINICAL TRIAL: NCT02848456
Title: The Effects of Spinal Manipulative Therapy on Postactivation Potentiation
Brief Title: The Effects of Spinal Manipulation on Central Nervous System Activity Measured by Reflexive Calf Muscle Recruitment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grant Sanders (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Grant Sanders, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-0507-F6A
Record Dates: First submitted 2016-07-13; First posted 2016-07-28 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Subluxation of Joint of Lumbar Spine
Keywords: Manipulation, Spinal; H-Reflex; Muscle Contraction; Muscle Strength Dynamometer
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Spinal Manipulation SM (Active Comparator): In a repeated measures, crossover design, all subjects received one of three randomized treatments during three separate sessions: SM; a 10 second plantar flexion maximal voluntary isometric contraction (MVIC) or the manipulation immediately preceding the contraction (SM+MVIC).
  Interventions: Procedure: Spinal Manipulation
- Max Voluntary Isometric Contraction MVIC (Active Comparator): In a repeated measures, crossover design, all subjects received one of three randomized treatments during three separate sessions: SM; a 10 second plantar flexion maximal voluntary isometric contraction (MVIC) or the manipulation immediately preceding the contraction (SM+MVIC).
  Interventions: Procedure: Max Voluntary Isometric Contraction
- SM+MVIC (Active Comparator): In a repeated measures, crossover design, all subjects received one of three randomized treatments during three separate sessions: SM; a 10 second plantar flexion maximal voluntary isometric contraction (MVIC) or the manipulation immediately preceding the contraction (SM+MVIC).
  Interventions: Procedure: SM+MVIC

INTERVENTIONS:
Procedure: Spinal Manipulation — Manual, side-posture, high-velocity low-amplitude spinal manipulation targeting the lower lumbar spine and sacroiliac joints
  Arms: Spinal Manipulation SM
Procedure: Max Voluntary Isometric Contraction — A 10 second plantar flexion maximal voluntary isometric contraction
  Arms: Max Voluntary Isometric Contraction MVIC
Procedure: SM+MVIC — The spinal manipulation immediately preceding the maximal voluntary isometric contraction
  Arms: SM+MVIC

SUMMARY:
This study investigated the effects of spinal manipulation on central nervous system activity. The presence of postactivation potentiation, an increase in muscular force production following prior muscular contractions, was measured with electromyography and the muscular force production during electrically-induced calf muscle reflexes. It was hypothesized that significantly greater potentiation would be stimulated by a calf muscle contraction with spinal manipulation delivered immediately beforehand than the potentiation arising from the contraction only.

DETAILED DESCRIPTION:
A randomized, controlled, single-blind crossover study design was utilized, and the three independent variables were spinal manipulative therapy (SMT), a 10 second plantar flexion maximal voluntary isometric contraction (MVIC) or SMT immediately preceding the MVIC (SMT + MVIC). The treatment order was randomized for each of the three sessions before the tibial nerve Hmax/Mmax stimulation protocol.

Each of the four dependent variables were evoked during the tibial nerve H-reflex stimulation protocol at the conclusion of each session, and included the Hmax/Mmax ratio (%) of the gastrocnemius and soleus muscles and the isometric twitch torque occurring at Hmax and at Mmax. Hmax, the highest H-reflex amplitude, is an indication of the greatest possible reflex activation; as such, it is an estimate of the number of motor neurons a subject is capable of activating in a given state. Further increases in the stimulation intensity cause the subsequent M-wave to reach its highest amplitude, Mmax. Mmax is a compound muscle action potential (CMAP) which represents full muscle activation. Specific to the current investigation, Mmax indicated activation of the total volume of the gastrocnemius/soleus motor neuron (MN) pool.

Given that Hmax is an inference of the number of MNs being recruited, and Mmax constitutes the entire motor neuron pool, the proportion of the entire MN pool capable of being recruited can be estimated with the Hmax/Mmax ratio. The Hmax/Mmax ratio was determined by division of the EMG peak-to-peak amplitudes (mV) evoked at Hmax by the preceding Mmax EMG peak-to-peak amplitudes. Differences in each of the four dependent variables (Hmax/Mmax ratios of the gastrocnemius and soleus and the peak twitch torques evoked at Hmax and Mmax) following each treatment form of SMT, MVIC or SMT+MVIC delivered during the three data collection sessions on three separate days were determined with a two-way (treatment × time point) repeated measures ANOVA. Percent changes from baseline were also calculated for each of the dependent variables, and the same type of ANOVA was used to determine differences in the within-subjects effects of each treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least one year of resistance training experience and current completion of at least three training sessions per week
* Males needed to be able to back squat a minimum load of 1.5 x body weight
* Females needed to be able to back squat 1 x body weight

Exclusion Criteria:

* Any pain in the lower back, abdomen or legs and/or surgeries performed in these regions

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in H-reflex amplitudes of the gastrocnemius and soleus muscles compared to baseline | Data were collected at 17 time points during a 20-minute tibial nerve electrical stimulation protocol post-treatment: 20 seconds, 40 seconds, 1:00, 2:00, 3:00, 4:00, 5:00, 6:00, 7:00, 8:00, 9:00, 10:00, 12:00, 14:00, 16:00, 18:00 and 20:00 minutes
  Peak-to-peak EMG amplitudes (mV) at Hmax of the gastrocnemius and soleus were recorded before and immediately following the three separate treatments
Changes in isometric twitch torques of the gastrocnemius and soleus muscles compared to baseline | Data were collected at 17 time points during a 20-minute tibial nerve electrical stimulation protocol post-treatment: 10 seconds, 30 seconds, 50 seconds, 1:30, 2:30, 3:30, 4:30, 5:30, 6:30, 7:30, 8:30, 9:30, 11:00, 13:00, 15:00, 17:00 and 19:00 minutes
  Twitch torques (Nm) of the gastrocnemius and soleus at Mmax were recorded before and immediately following the three separate treatments

CONTACTS AND LOCATIONS:
Overall Officials: Grant D Sanders, D.C., Ph.D., Principal Investigator — College of Education, Department of Kinesiology and Health Promotion, University of Kentucky, Lexington, KY; James W Yates, Ph.D., Study Chair — College of Education, Department of Kinesiology and Health Promotion, University of Kentucky, Lexington, KY
Locations (1):
- College of Education, Department of Kinesiology and Health Promotion, University of Kentucky, Lexington, KY, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Shared data include the subjects' reflexive EMG amplitudes and peak torques of the gastrocnemius and soleus during the Hoffmann Reflex electrical stimulation protocol at the conclusion of each data collection session. These raw data are available in Appendix K of the PI's dissertation, which may be obtained at http://uknowledge.uky.edu/khp_etds/27/

REFERENCES:
- [Background] Hurwitz EL. Epidemiology: spinal manipulation utilization. J Electromyogr Kinesiol. 2012 Oct;22(5):648-54. doi: 10.1016/j.jelekin.2012.01.006. Epub 2012 Jan 29. PMID 22289432
- [Background] Michaleff ZA, Lin CW, Maher CG, van Tulder MW. Spinal manipulation epidemiology: systematic review of cost effectiveness studies. J Electromyogr Kinesiol. 2012 Oct;22(5):655-62. doi: 10.1016/j.jelekin.2012.02.011. Epub 2012 Mar 18. PMID 22429823
- [Background] Goertz CM, Long CR, Hondras MA, Petri R, Delgado R, Lawrence DJ, Owens EF, Meeker WC. Adding chiropractic manipulative therapy to standard medical care for patients with acute low back pain: results of a pragmatic randomized comparative effectiveness study. Spine (Phila Pa 1976). 2013 Apr 15;38(8):627-34. doi: 10.1097/BRS.0b013e31827733e7. PMID 23060056
- [Background] Goertz CM, Pohlman KA, Vining RD, Brantingham JW, Long CR. Patient-centered outcomes of high-velocity, low-amplitude spinal manipulation for low back pain: a systematic review. J Electromyogr Kinesiol. 2012 Oct;22(5):670-91. doi: 10.1016/j.jelekin.2012.03.006. Epub 2012 Apr 24. PMID 22534288
- [Background] von Heymann WJ, Schloemer P, Timm J, Muehlbauer B. Spinal high-velocity low amplitude manipulation in acute nonspecific low back pain: a double-blinded randomized controlled trial in comparison with diclofenac and placebo. Spine (Phila Pa 1976). 2013 Apr 1;38(7):540-8. doi: 10.1097/BRS.0b013e318275d09c. PMID 23026869
- [Background] Boline PD, Kassak K, Bronfort G, Nelson C, Anderson AV. Spinal manipulation vs. amitriptyline for the treatment of chronic tension-type headaches: a randomized clinical trial. J Manipulative Physiol Ther. 1995 Mar-Apr;18(3):148-54. PMID 7790794
- [Background] Nelson CF, Bronfort G, Evans R, Boline P, Goldsmith C, Anderson AV. The efficacy of spinal manipulation, amitriptyline and the combination of both therapies for the prophylaxis of migraine headache. J Manipulative Physiol Ther. 1998 Oct;21(8):511-9. PMID 9798179
- [Background] Burton AK, Tillotson KM, Cleary J. Single-blind randomised controlled trial of chemonucleolysis and manipulation in the treatment of symptomatic lumbar disc herniation. Eur Spine J. 2000 Jun;9(3):202-7. doi: 10.1007/s005869900113. PMID 10905437
- [Background] Haas M, Sharma R, Stano M. Cost-effectiveness of medical and chiropractic care for acute and chronic low back pain. J Manipulative Physiol Ther. 2005 Oct;28(8):555-63. doi: 10.1016/j.jmpt.2005.08.006. PMID 16226622
- [Background] Korthals-de Bos IB, Hoving JL, van Tulder MW, Rutten-van Molken MP, Ader HJ, de Vet HC, Koes BW, Vondeling H, Bouter LM. Cost effectiveness of physiotherapy, manual therapy, and general practitioner care for neck pain: economic evaluation alongside a randomised controlled trial. BMJ. 2003 Apr 26;326(7395):911. doi: 10.1136/bmj.326.7395.911. PMID 12714472
- [Background] Gunnar Brolinson P, McGinley SM, Kerger S. Osteopathic manipulative medicine and the athlete. Curr Sports Med Rep. 2008 Feb;7(1):49-56. doi: 10.1097/01.CSMR.0000308664.13278.a7. PMID 18296946
- [Background] Julian C, Hoskins W, Vitiello AL. Sports chiropractic management at the World Ice Hockey Championships. Chiropr Osteopat. 2010 Dec 3;18:32. doi: 10.1186/1746-1340-18-32. PMID 21129212
- [Background] Nook DD, Nook BC. A report of the 2009 World Games injury surveillance of individuals who voluntarily used the International Federation of Sports Chiropractic delegation. J Manipulative Physiol Ther. 2011 Jan;34(1):54-61. doi: 10.1016/j.jmpt.2010.11.003. PMID 21237408
- [Background] Uchacz GP. 2010 olympic winter games chiropractic: the making of history. J Can Chiropr Assoc. 2010 Mar;54(1):14-6. No abstract available. PMID 20195421
- [Background] Miners AL. Chiropractic treatment and the enhancement of sport performance: a narrative literature review. J Can Chiropr Assoc. 2010 Dec;54(4):210-21. PMID 21120012
- [Background] Robbins DW. Postactivation potentiation and its practical applicability: a brief review. J Strength Cond Res. 2005 May;19(2):453-8. doi: 10.1519/R-14653.1. PMID 15903390
- [Background] Wilson JM, Duncan NM, Marin PJ, Brown LE, Loenneke JP, Wilson SM, Jo E, Lowery RP, Ugrinowitsch C. Meta-analysis of postactivation potentiation and power: effects of conditioning activity, volume, gender, rest periods, and training status. J Strength Cond Res. 2013 Mar;27(3):854-9. doi: 10.1519/JSC.0b013e31825c2bdb. PMID 22580978
- [Background] Gouvea AL, Fernandes IA, Cesar EP, Silva WA, Gomes PS. The effects of rest intervals on jumping performance: a meta-analysis on post-activation potentiation studies. J Sports Sci. 2013;31(5):459-67. doi: 10.1080/02640414.2012.738924. Epub 2012 Nov 9. PMID 23140550
- [Background] Hodgson M, Docherty D, Robbins D. Post-activation potentiation: underlying physiology and implications for motor performance. Sports Med. 2005;35(7):585-95. doi: 10.2165/00007256-200535070-00004. PMID 16026172
- [Background] Tillin NA, Bishop D. Factors modulating post-activation potentiation and its effect on performance of subsequent explosive activities. Sports Med. 2009;39(2):147-66. doi: 10.2165/00007256-200939020-00004. PMID 19203135
- [Background] Sale DG. Postactivation potentiation: role in human performance. Exerc Sport Sci Rev. 2002 Jul;30(3):138-43. doi: 10.1097/00003677-200207000-00008. PMID 12150573
- [Background] Hamada T, Sale DG, MacDougall JD, Tarnopolsky MA. Postactivation potentiation, fiber type, and twitch contraction time in human knee extensor muscles. J Appl Physiol (1985). 2000 Jun;88(6):2131-7. doi: 10.1152/jappl.2000.88.6.2131. PMID 10846027
- [Background] Chiu LZ, Fry AC, Weiss LW, Schilling BK, Brown LE, Smith SL. Postactivation potentiation response in athletic and recreationally trained individuals. J Strength Cond Res. 2003 Nov;17(4):671-7. doi: 10.1519/1533-4287(2003)0172.0.co;2. PMID 14636093
- [Background] Lorenz D. Postactivation potentiation: an introduction. Int J Sports Phys Ther. 2011 Sep;6(3):234-40. PMID 21904700
- [Background] Palmieri RM, Ingersoll CD, Hoffman MA. The hoffmann reflex: methodologic considerations and applications for use in sports medicine and athletic training research. J Athl Train. 2004 Jul;39(3):268-77. PMID 16558683
- [Background] Knikou M. The H-reflex as a probe: pathways and pitfalls. J Neurosci Methods. 2008 Jun 15;171(1):1-12. doi: 10.1016/j.jneumeth.2008.02.012. Epub 2008 Mar 4. PMID 18394711
- [Background] Comyns TM, Harrison AJ, Hennessy L, Jensen RL. Identifying the optimal resistive load for complex training in male rugby players. Sports Biomech. 2007 Jan;6(1):59-70. doi: 10.1080/14763140601058540. PMID 17542178
- [Background] Thompsen AG, Kackley T, Palumbo MA, Faigenbaum AD. Acute effects of different warm-up protocols with and without a weighted vest on jumping performance in athletic women. J Strength Cond Res. 2007 Feb;21(1):52-6. doi: 10.1519/00124278-200702000-00010. PMID 17313270
- [Background] Zehr EP. Considerations for use of the Hoffmann reflex in exercise studies. Eur J Appl Physiol. 2002 Apr;86(6):455-68. doi: 10.1007/s00421-002-0577-5. Epub 2002 Mar 7. PMID 11944092
- [Background] Folland JP, Wakamatsu T, Fimland MS. The influence of maximal isometric activity on twitch and H-reflex potentiation, and quadriceps femoris performance. Eur J Appl Physiol. 2008 Nov;104(4):739-48. doi: 10.1007/s00421-008-0823-6. Epub 2008 Jul 30. PMID 18665389
- [Background] Pickar JG, Kang YM. Paraspinal muscle spindle responses to the duration of a spinal manipulation under force control. J Manipulative Physiol Ther. 2006 Jan;29(1):22-31. doi: 10.1016/j.jmpt.2005.11.014. PMID 16396726
- [Background] Mitchell CJ, Sale DG. Enhancement of jump performance after a 5-RM squat is associated with postactivation potentiation. Eur J Appl Physiol. 2011 Aug;111(8):1957-63. doi: 10.1007/s00421-010-1823-x. Epub 2011 Jan 13. PMID 21229259
- [Background] Rixon KP, Lamont HS, Bemben MG. Influence of type of muscle contraction, gender, and lifting experience on postactivation potentiation performance. J Strength Cond Res. 2007 May;21(2):500-5. doi: 10.1519/R-18855.1. PMID 17530946
- [Background] McNeil CJ, Butler JE, Taylor JL, Gandevia SC. Testing the excitability of human motoneurons. Front Hum Neurosci. 2013 Apr 24;7:152. doi: 10.3389/fnhum.2013.00152. eCollection 2013. PMID 23630483
- [Background] Gossen ER, Sale DG. Effect of postactivation potentiation on dynamic knee extension performance. Eur J Appl Physiol. 2000 Dec;83(6):524-30. doi: 10.1007/s004210000304. PMID 11192060
- [Background] Hodgson MJ, Docherty D, Zehr EP. Postactivation potentiation of force is independent of h-reflex excitability. Int J Sports Physiol Perform. 2008 Jun;3(2):219-31. doi: 10.1123/ijspp.3.2.219. PMID 19208930
- [Background] Enoka RM, Hutton RS, Eldred E. Changes in excitability of tendon tap and Hoffmann reflexes following voluntary contractions. Electroencephalogr Clin Neurophysiol. 1980 Jun;48(6):664-72. doi: 10.1016/0013-4694(80)90423-x. PMID 6155255
- [Background] Hoch MC, Krause BA. Intersession reliability of H:M ratio is greater than the H-reflex at a percentage of M-max. Int J Neurosci. 2009;119(3):345-52. doi: 10.1080/00207450802480309. PMID 19116841
- [Background] Pickar JG, Sung PS, Kang YM, Ge W. Response of lumbar paraspinal muscles spindles is greater to spinal manipulative loading compared with slower loading under length control. Spine J. 2007 Sep-Oct;7(5):583-95. doi: 10.1016/j.spinee.2006.10.006. Epub 2007 Jan 10. PMID 17905321
- [Background] Dishman JD, Bulbulian R. Spinal reflex attenuation associated with spinal manipulation. Spine (Phila Pa 1976). 2000 Oct 1;25(19):2519-24;discussion 2525. doi: 10.1097/00007632-200010010-00015. PMID 11013505
- [Background] Dishman JD, Bulbulian R. Comparison of effects of spinal manipulation and massage on motoneuron excitability. Electromyogr Clin Neurophysiol. 2001 Mar;41(2):97-106. PMID 11284061
- [Background] Dishman JD, Ball KA, Burke J. First Prize: Central motor excitability changes after spinal manipulation: a transcranial magnetic stimulation study. J Manipulative Physiol Ther. 2002 Jan;25(1):1-9. PMID 11898013
- [Background] Dishman JD, Burke J. Spinal reflex excitability changes after cervical and lumbar spinal manipulation: a comparative study. Spine J. 2003 May-Jun;3(3):204-12. doi: 10.1016/s1529-9430(02)00587-9. PMID 14589201
- [Background] Dishman JD, Dougherty PE, Burke JR. Evaluation of the effect of postural perturbation on motoneuronal activity following various methods of lumbar spinal manipulation. Spine J. 2005 Nov-Dec;5(6):650-9. doi: 10.1016/j.spinee.2005.08.007. PMID 16291107
- [Background] Dishman JD, Weber KA 2nd, Corbin RL, Burke JR. Understanding inhibitory mechanisms of lumbar spinal manipulation using H-reflex and F-wave responses: a methodological approach. J Neurosci Methods. 2012 Sep 30;210(2):169-77. doi: 10.1016/j.jneumeth.2012.07.014. Epub 2012 Jul 31. PMID 22878176
- [Background] Fryer G, Pearce AJ. The effect of lumbosacral manipulation on corticospinal and spinal reflex excitability on asymptomatic participants. J Manipulative Physiol Ther. 2012 Feb;35(2):86-93. doi: 10.1016/j.jmpt.2011.09.010. Epub 2011 Oct 28. PMID 22036580
- [Background] Patikas DA, Bassa H, Kotzamanidis C. Changes in the reflex excitability during and after a sustained, low-intensity muscle contraction. Int J Sports Med. 2006 Feb;27(2):124-30. doi: 10.1055/s-2005-837490. PMID 16475058
- [Background] Trimble MH, Harp SS. Postexercise potentiation of the H-reflex in humans. Med Sci Sports Exerc. 1998 Jun;30(6):933-41. doi: 10.1097/00005768-199806000-00024. PMID 9624654